CLINICAL TRIAL: NCT01109186
Title: Role of Specific Immune Cellular Response in the Control of BK Virus Infection: Prospective Study, Monocentric and Longitudinal During the First Nine Months After a Kidney Transplantation
Brief Title: Anti-BK Virus Immune Response and Kidney Transplantation
Acronym: BKv
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: BRD/10/03-ZF
Record Dates: First submitted 2010-04-21; First posted 2010-04-23 (Estimated); Last update posted 2021-09-17 (Actual); Status verified 2021-09

CONDITIONS: Kidney Transplantation
Keywords: patient with a kidney transplantation since less than 30 days

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- kidney-transplanted patients
  Interventions: Other: biological parameters

INTERVENTIONS:
Other: biological parameters — blood sample at M1, M2, M3; M4; M5, M6, M7, M8 and M9 after kidney transplantation

SUMMARY:
BK virus infections are very frequent during months following a kidney transplantation: a viral reactivation is observed for almost 50% of patients during first year. This reactivation leads to a viremia for 10 to 15% of patient during this same period. The most frequent complication is interstitial nephritis for 2 to 8% of patients (27 patients representing 2.7% during 6 years in Nantes).

An intensive et persisting viral replication, assessed by detection of high blood viral load, could evolved to a viral nephropathy which lead to a very pejorative functional issue for the graft.

Biological follow-up of these infections lay on the measures of viral load. Their positivity must alert the physician and lead him to modulate immunosuppressive treatment.

Actually, there is no real consensus about the modalities of pharmacological immunosuppression decrease (decrease dose or change of molecule).

Specific lymphocytic anti-BKv evaluated on several cohorts of patients permit to prove:

* weakness of immune cellular response for patient with high viremia
* increase of this response when viral load decrease These studies laid on detection of INFg synthesis by Elispot after stimulation with viral antigens and in vitro cellular expansion.

New prospective and longitudinal data comparing the immune cellular response (systematic and early) after graft between patients controlling or not BKv infection are necessary to improve the comprehension of illness natural history.

The investigators propose to enlarge the investigation of anti-BKv immune cellular response to other functions than IFNg synthesis in the aim of detecting the eventual role of polyfunctional lymphocytes for infection control. Furthermore, the investigators propose to identify better diagnostic and prognostic makers.

ELIGIBILITY:
Inclusion Criteria:

* Kidney-transplanted patient, since less than 30 days
* Older than 18 years old
* Treatment with tacrolimus and mycophénolate mofetil

Exclusion Criteria:

* No informed consent
* Pregnant women
* Patient under legal guardianship
* Treated by ciclosporin or mTOR-inhibitor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Kidney-transplanted person
Sampling Method: Non-Probability Sample
Enrollment: 158 (Actual)
Dates: Start 2010-11-30 (Actual); Primary Completion 2014-08-26 (Actual); Study Completion 2015-09-01 (Actual)

PRIMARY OUTCOMES:
Comparison of the level of response between patient with a "non-controlled infection" and patients for who the blood viral load is under 103 copBKv/ml. | at 1month, 2months, 3months, 4, 5, 6, 7, 8 and 9 months after kidney transplantation
  Analyse the role of T-lymphocytes response in the control of BKv infection

SECONDARY OUTCOMES:
Analyse of the other causes that could influence the occurence of a viremia higher than 103 copBKv/ml | at 1month, 2months, 3months, 4, 5, 6, 7, 8 and 9 months after kidney transplantation
  Other causes for abnormal viremia
Measurement of histological consequences of a BKv non-controlled infection during the first year post-graft | at 12 months after kidney transplantation
  Determine the frequence of occurence of nephropathy due to BKv for the population with a non-controlled infection
Measurement of increase of immune response due to modifications of immunosuppressive treatment for patient with a non-controlled infection | at 1, 3 et 6 months after modification of immunosuppressive treatment
  Comparision between the level of immune response and the time when the first viremia is higher than 103 copBKv/ml and 1, 3 et 6 months after modification of immunosuppressive treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Nantes' Univeristy hospital, Nantes, France